CLINICAL TRIAL: NCT01110187
Title: A Pilot Study of NSICU Assessment of Seizure Prophylaxis With Lacosamide
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollement
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Jerzy P Szaflarski, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JPS-001
Record Dates: First submitted 2010-04-16; First posted 2010-04-26 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-02

CONDITIONS: Traumatic Brain Injury
Keywords: Lacosamide; Fosphenytoin; traumatic brain injury; Glasgow coma scale; Disability Rating Scale; Resource Utilization Questionnaire; Continuous EEG; seizures
MeSH Terms: conditions — Brain Injuries, Traumatic; Seizures | interventions — Lacosamide; fosphenytoin; Phenytoin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV LCM (lacosamide) (Experimental): Patients with severe traumatic brain injury (TBI) or subarachanoid hemorrhage (SAH) randomized to seizure prophylaxis with either lacosamide.
  Interventions: Drug: lacosamide
- IV fPHT (fos-phenytoin) (Active Comparator): Patients with TBI or SAH randomized to seizure prophylaxis with fos-phenytoin
  Interventions: Drug: Fosphenytoin

INTERVENTIONS:
Drug: lacosamide — 200 mg IV over 60 minutes; these patients will then be started on a maintenance dose 100 mg, IV BID as prophylaxis administered as per pharmacy protocol consistent with acceptable standards of care for 7 days. The Lacosamide dose can be adjusted as needed if seizures occur for therapeutic effect up to 200 mg bid (400 mg/d) as a maximum dose.
  Other Names: Vimpat
  Arms: IV LCM (lacosamide)
Drug: Fosphenytoin — 20 mgPE/kg IV over 60 minutes and then will be started on a maintenance dose (5 mgPE/kg/day, rounded to nearest dose of 150 mgPE IV, BID administered as per pharmacy protocol consistent with acceptable standards of care for 7 days
  Other Names: Dilantin
  Arms: IV fPHT (fos-phenytoin)

SUMMARY:
Trial to determine if seizure prophylaxis with IV LCM in NSICU patients experiencing mental status changes due to severe traumatic brain injury (sTBI) will result in improved short- and long-term outcomes and better immediate adverse effects when compared to the current standard of care anticonvulsant (IV fPHT) and will be at least as effective as IV fPHT in preventing clinical and sub-clinical seizure activity.

DETAILED DESCRIPTION:
The goals are to compare IV LCM and IV fPHT for seizure prophylaxis in the neuro-critical care setting in terms of the following outcome measures:

1. The short- and long-term incidence of adverse events related to the anticonvulsant medication
2. The frequency of clinically-evident and sub-clinical seizures, as demonstrated by continuous EEG monitoring for the first three days and by clinical assessment for up to 6 months after initial admission.
3. Intermediate and long-term outcomes as measured by standard outcome measures including Extended Glasgow Outcome Scale, Disability Rating Scale, and Resource Utilization Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Subject with traumatic brain injury admitted to the hospital less than 24 hours prior to randomization
* GCS score 3-8 (inclusive) or GCS motor score of 5 or less and abnormal admission CT scan showing intracranial pathology
* Hemodynamically stable with a systolic BP > 90 mmHg
* At least one reactive pupil
* Age at least 18 years
* Signed informed consent and HIPAA authorization for research form
* Patients will not be excluded because of race, gender, educational status or occupation

Exclusion Criteria:

* No venous access
* Spinal cord injury
* History of or CT confirmation of previous brain injury such as brain tumor, cerebral infarct, or spontaneous intracerebral hemorrhage
* Hemodynamically unstable
* Suspected anoxic events
* Other peripheral trauma likely to result in liver failure
* Age less than 18 years of age
* Known hypersensitivity to any anticonvulsant
* Any treatment, condition, or injury that contraindicates treatment with Lacosamide (LCM) or fos-phenytoin (fPHT)
* Inability to obtain signed informed consent or HIPAA authorization for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy P Szaflarski, M.D., PhD, Principal Investigator — Univeristy of Cincinnati
Locations (3):
- United States (3):
  - UC Health University Pointe, Cincinnati, Ohio
  - UC Health Medical Arts Building, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio

REFERENCES:
- [Background] Szaflarski JP, Sangha KS, Lindsell CJ, Shutter LA. Prospective, randomized, single-blinded comparative trial of intravenous levetiracetam versus phenytoin for seizure prophylaxis. Neurocrit Care. 2010 Apr;12(2):165-72. doi: 10.1007/s12028-009-9304-y. PMID 19898966

RESULTS

PARTICIPANT FLOW:
Groups:
- IV LCM: Patients with severe TBI later randomized to seizure prophylaxis with LCM (Lacosamide). For IV LCM dosing and adjustment see "Intervention" section.
- IV fPHT: Patients randomized to fPHT (fos-phenytoin) with moderate or severe TBI. For IV fPHT dosing and adjustment see "Intervention" section.
Period: Overall Study
Arm/Group | IV LCM | IV fPHT
Started | 7 | 4
Completed | 7 (completed 7 day treatment) | 4 (completed 7 day treatment)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Traumatic Brain Injury
Groups:
- IV LCM: patients randomized to IV LCM (7)
- IV fPHT: patients randomized to IV fPHT (4)
- Total: Total of all reporting groups
Arm/Group | IV LCM | IV fPHT | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 66] | 55.5 [23 to 61] | 56 [23 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The primary outcome measure is the incidence of clinical adverse events. These will be followed by daily clinical observations during the hospital stay. Subjects will be evaluated for e.g., seizures, fever, neurological changes, cardiovascular, hematologic and dermatologic abnormalities, liver failure, renal failure, and death; EKGs will be requested as per ICU routines through day 7.
Time Frame: baseline to 7 days
Population: all participants in each arm were available for analyses
Measure: Number; unit: number of events experienced
Groups:
- IV LCM: Patients with severe TBI later randomized to seizure prophylaxis with lacosamide.
- IV fPHT: Patients with severe TBI randomized to seizure prophylaxis with fPHT
Arm/Group | IV LCM | IV fPHT
Number analyzed (Participants) | 7 | 4
number of events experienced | 12 | 21

2. Secondary Outcome: Number of Participants With Seizures
Description: Number of seizures in the first 72 hours based on EEG recording
Time Frame: baseline to 72 hours
Measure: Number; unit: number of participants with seizures
Groups:
- IV LCM: Patients with severe traumatic brain injury (TBI) or subarachanoid hemorrhage (SAH) randomized to seizure prophylaxis with either lacosamide.
  lacosamide: 200 mg IV over 60 minutes; these patients will then be started on a maintenance dose 100 mg, IV BID as prophylaxis administered as per pharmacy protocol consistent with acceptable standards of care for 7 days. The Lacosamide dose can be adjusted as needed if seizures occur for therapeutic effect up to 200 mg bid (400 mg/d) as a maximum dose.
- IV fPHT: Patients with TBI or SAH randomized to seizure prophylaxis with fos-phenytoin
  Fosphenytoin: 20 mgPE/kg IV over 60 minutes and then will be started on a maintenance dose (5 mgPE/kg/day, rounded to nearest dose of 150 mgPE IV, BID administered as per pharmacy protocol consistent with acceptable standards of care for 7 days
Arm/Group | IV LCM | IV fPHT
Number analyzed (Participants) | 7 | 4
number of participants with seizures | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline to 7 days
Groups:
- IV fPHT: Patients with severe TBI later randomized to seizure prophylaxis with phenytoin.
Arm/Group | IV LCM | IV fPHT
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV LCM (N=7) | IV fPHT (N=4)
death (Nervous system disorders) | 2 (2) | 0 (0) — death because of baseline condition (TBI) - expected
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV LCM (N=7) | IV fPHT (N=4)
fever (Investigations) | 3 (3) | 3 (3)
increased ICP (Nervous system disorders) | 0 (0) | 3 (3)
Hypotension (Investigations) | 0 (0) | 1 (1)
LFT (Hepatobiliary disorders) | 1 (1) | 3 (3)
stroke (Nervous system disorders) | 1 (1) | 3 (3)
arrythmia (Cardiac disorders) | 1 (1) | 3 (3)
anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
low platelets (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to lack of enrollment. Statistical comparisons between groups are not possible and were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No